CLINICAL TRIAL: NCT02961361
Title: the Effect of Dexmedetomidine in Coracoid Approach Brachial Plexus Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dex
Record Dates: First submitted 2016-10-22; First posted 2016-11-11 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Injury of Upper Limb
Keywords: dexmedetomidine; coracoid; brachial plexus block
MeSH Terms: conditions — Arm Injuries | interventions — Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Control (Experimental): 40 ml 0.375% ropivacaine was injected after Locating brachial plexus.
  Interventions: Drug: ropivacaine
- Group Dexmedetomidine (Experimental): 40 ml 0.375% ropivacaine mixed with dexmedetomidine was injected after Locating brachial plexus.
  Interventions: Drug: ropivacaine mixed with dexmedetomidine

INTERVENTIONS:
Drug: ropivacaine — 40 ml 0.375% ropivacaine was injected after Locating brachial plexus.
  Arms: Group Control
Drug: ropivacaine mixed with dexmedetomidine — 40 ml 0.375% ropivacaine mixed with dexmedetomidine was injected after Locating brachial plexus.
  Arms: Group Dexmedetomidine

SUMMARY:
Dexmedetomidine is an α-2 adrenoreceptor agonist and has been extensively used through intravenous infusion，in order to improved the quality of block in regional anesthesia. In this prospective, randomized study, the authors focus on the effect of dexmedetomidine mixed with ropivacaine in coracoid approach brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status I or II;
2. Aged 18-60 years;
3. The elbow, forearm, wrist or hand surgery

Exclusion Criteria:

1. History of allergy to local anesthetics;
2. Coagulation dysfunction, neuromuscular disease or local infection;
3. The operation time is longer than the local anesthetics effective time.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-12 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
duration time | once per hour after surgery until 24 hours after surgery
  effective analgesia time

SECONDARY OUTCOMES:
onset time | 5,10,15,20,25,30 min after injection
Visual analogue scale | 2,6,12,24hour after injection

CONTACTS AND LOCATIONS:
Overall Officials: wensheng he, MD, Principal Investigator — Hebei Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He WS, Liu Z, Wu ZY, Sun HJ, Yang XC, Wang XL. The effect of dexmedetomidine in coracoid approach brachial plexus block under dual stimulation. Medicine (Baltimore). 2018 Sep;97(39):e12240. doi: 10.1097/MD.0000000000012240. PMID 30278495